CLINICAL TRIAL: NCT02086578
Title: Phase II Study Assessing the Potential for Reduced Rates of Implant Failure Using Multi-Beam Intensity-Modulated Radiation Therapy for Locally Advanced Breast Cancer Patients With Implant Reconstructions
Brief Title: Study Assessing the Potential for Reduced Rates of Implant Failure Using Multi-Beam Intensity-Modulated Radiation Therapy for Locally Advanced Breast Cancer Patients With Implant Reconstructions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-028
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: multi-beam Intensity-Modulated Radiation Therapy (IMRT); 14-028
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- Group 1 (Experimental): Physical examination by MD, optional Breast MRI, Breast-Q© at baseline (after permanent implant exchange, physical exam and Breast-Q© may be done after the initiation of IMRT), 12 ± 2 months and 24 ± 2 months post- IMRT. Total length of the follow-up time will be 24 ± 2 months post-IMRT. A subset of 10 left-sided patients will receive 13N-NH3 PET scans within the radiation simulation session. A CT for coronary calcium scoring and a low-dose CT for attenuation correction will also be obtained at this time. Myocardial blood flow will be measured during rest and at peak stress with 13N-NH3 as a perfusion tracer. A follow-up 13N-NH3 PET study with low-dose CT for attenuation correction will be obtained 12-18 months (± 6 months) post-IMRT.
  Interventions: Device: Breast MRI; Behavioral: Breast-Q© questionnaire; Radiation: Multi-Beam IMRT
- Group 2 (Experimental): Physical examination by MD, optional Breast MRI, Breast-Q © at baseline (after permanent implant exchange and after IMRT), 18 ± 2 months and 30 ± 2 months post-IMRT, as these patients will undergo exchange of the temporary expander for the permanent implant approximately 4-8 months following the completion of radiation (at the discretion of the treating plastic surgeon). Total length of the follow-up time will be 30 ± 2 months post-IMRT
  Interventions: Device: Breast MRI; Behavioral: Breast-Q© questionnaire; Radiation: Multi-Beam IMRT

INTERVENTIONS:
Device: Breast MRI
Behavioral: Breast-Q© questionnaire
Radiation: Multi-Beam IMRT — The radiation dose (50-50.4 Gy/25-28 fractions in approximately 5-6 weeks), treatment-planning and delivery aspects are according to departmental guidelines for breast IMRT.

SUMMARY:
The purpose of this study is to determine if a radiation treatment called "Multi-beam Intensity Modulated Radiation Therapy"(IMRT) can reduce side effects related to your implant if they are a candidate for radiation therapy. Currently, the standard method of giving radiation is with "3D radiation", which only uses 2-5 beams of radiation. "Multi-beam" IMRT works by using 8-12 small radiation beams to give a more "tailored" or "customized" radiation dose to the implant, breast, chest wall and lymph nodes. At the same time, multi-beam IMRT may lower the radiation dose to the heart, lung and nearby tissues. The goal of the study is to reduce complications after irradiation to the implants.

The study doctors have recently completed a trial using this technique and are now specifically looking at its impact on women with implant reconstructions who are undergoing post-mastectomy radiation therapy. By delivering a more "customized" dose of radiation to the implant, the intent is to reduce side effects of radiation on the implant.

DETAILED DESCRIPTION:
Patients will undergo mastectomy and axillary dissection with immediate tissue expander placement. As is the current practice at MSKCC, patients receiving adjuvant chemotherapy will undergo expansion during chemotherapy, with exchange for a permanent implant to be performed approximately one month after chemotherapy and radiation to begin approximately one month after exchange. Patients who receive neoadjuvant chemotherapy will undergo "rapid expansion" of the expander and begin radiation at least 4 weeks following surgery, although it may be performed sooner if the patient has recovered from surgery and the treating physician deems it safe to proceed with treatment. In these patients, exchange for the permanent implant will occur at the discretion of the treating plastic surgeon (approximately 5-8 months after the end of radiation).

ELIGIBILITY:
Inclusion Criteria:

* Females who are age ≥ 18 years of age with a life expectancy estimated to be at least 2 years
* Histologically-confirmed invasive breast cancer by MSKCC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Status post mastectomy with surgical assessment of axillary nodes
* Immediate reconstruction with tissue expander (Group 2) or permanent implant (Group 1) prior to RT performed at MSKCC
* If PMRT is recommended, the treatment fields will include the axillary, supraclavicular, and internal mammary nodes.

Exclusion Criteria:

* Absence of a breast reconstruction prior to RT (placement of tissue expander is sufficient for group 2)
* Pregnant or breastfeeding.
* Psychiatric or addictive disorders that would preclude obtaining informed consent or filling out Breast-Q© questionnaires.
* Prior radiation therapy to the ipsilateral breast/nodes or thorax.
* The criterias outlined above apply to the patients enrolled to meet the primary objective of the study. Additional criteria for patients in the cardiac substudy portion of the protocol are outlined in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daphna Gelblum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Follow-Up only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- IMRT to Temporary Expander: Physical examination by MD, optional Breast MRI, Breast-Q© at baseline (after permanent implant exchange, physical exam and Breast-Q© may be done after the initiation of IMRT), 12 ± 2 months and 24 ± 2 months post- IMRT. Total length of the follow-up time will be 24 ± 2 months post-IMRT. A subset of 10 left-sided patients will receive 13N-NH3 PET scans within the radiation simulation session. A CT for coronary calcium scoring and a low-dose CT for attenuation correction will also be obtained at this time. Myocardial blood flow will be measured during rest and at peak stress with 13N-NH3 as a perfusion tracer. A follow-up 13N-NH3 PET study with low-dose CT for attenuation correction will be obtained 12-18 months (± 6 months) post-IMRT.
  Breast MRI
  Breast-Q© questionnaire
  Multi-Beam IMRT: The radiation dose (50-50.4 Gy/25-28 fractions in approximately 5-6 weeks), treatment-planning and delivery aspects are according to departmental guidelines for breast IMRT.
- IMRT to Permanent Implant: Physical examination by MD, optional Breast MRI, Breast-Q © at baseline (after permanent implant exchange and after IMRT), 18 ± 2 months and 30 ± 2 months post-IMRT, as these patients will undergo exchange of the temporary expander for the permanent implant approximately 4-8 months following the completion of radiation (at the discretion of the treating plastic surgeon). Total length of the follow-up time will be 30 ± 2 months post-IMRT
  Breast MRI
  Breast-Q© questionnaire
  Multi-Beam IMRT: The radiation dose (50-50.4 Gy/25-28 fractions in approximately 5-6 weeks), treatment-planning and delivery aspects are according to departmental guidelines for breast IMRT.
Period: Overall Study
Arm/Group | IMRT to Temporary Expander | IMRT to Permanent Implant
Started | 42 | 58
Completed | 42 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes participants who were able to complete study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMRT to Temporary Expander | IMRT to Permanent Implant | Total
Number analyzed (Participants) | 42 | 58 | 100
Age, Continuous [Median (Full Range); unit: years] | 56 [46 to 60] | 54 [46 to 64] | 54 [46 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 58 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 40 | 53 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 8 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 30 | 39 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 58 | 100

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Implant Failure
Description: The multi-beam IMRT would be considered efficacious if the incidence of implant failure is reduced by at least a relative 30% by the end of the study period (24 months post-IMRT for Group 1, and 30 months post-IMRT for Group 2).
Time Frame: 24 months post-IMRT for Group 1, and 30 months post-IMRT for Group 2
Measure: Number; unit: Number of Participants with Implant Fail
Arm/Group | IMRT to Temporary Expander | IMRT to Permanent Implant
Number analyzed (Participants) | 42 | 58
Number of Participants with Implant Fail
  Implant Failure | 8 | 17
  No Implant Failure | 34 | 41

2. Secondary Outcome: Incidence of Moderate to Severe Capsular Contracture
Description: Will be examined using number of participants who developed Baker's grade <2 and ≥2 capsular contracture, respectively, at 12 or 18 months and 24 or 30 months after IMRT was administered. Participants were assigned a Baker Classification score (a standardized 4-point scale, which integrates the texture and appearance of the breast) at baseline and each follow-up interval by the radiation oncologist or plastic surgeon (the higher of the 2 was used if the score was discordant). Significant capsular contracture is measured as Baker grade III or IV.
Time Frame: 24 months post-IMRT for Group 1, and 30 months post-IMRT for Group 2
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT to Temporary Expander | IMRT to Permanent Implant
Number analyzed (Participants) | 42 | 58
Participants
  Grade IA-II Capsular Contracture | 26 | 36
  Grade III-IV Capsular Contracture | 16 | 11
  No Capsular Contracture | 0 | 11

3. Secondary Outcome: Rates of Minor Revisional Surgeries
Description: Incidence of minor revisional surgeries by plastic surgeon will be evaluated by proportions too. Again, the rates (proportions) will be compared across the two groups.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT to Temporary Expander | IMRT to Permanent Implant
Number analyzed (Participants) | 42 | 58
Participants
  Participants with minor surgical corrections | 0 | 2
  Participants without minor surgical corrections | 42 | 56

4. Secondary Outcome: Evaluate Cosmesis
Description: To evaluate cosmesis, the Breast-Q© will be utilized in these assessments and will be presented descriptively, giving summary statistics for changes in the Breast-Q© scores over time. With a focus on the post-operative period, the module will evaluate changes over time in four of the six subthemes identified by Breast-Q: (1) Psychosocial well-being; (2) Physical well-being; (3) Satisfaction with breasts; and (4) Satisfaction with outcome. Each subtheme will be evaluated using one or more scales. Each scale is independently scored into a value that ranges from 0 to 100, with higher score indicating greater satisfaction or better health-related quality of life.
Time Frame: Baseline, Follow-up 1 (Arm 1:12 months (± 2 mo); Arm 2:12-18 months (± 6 mo)), Follow-up 2 (Arm 1:12-18 months (± 6 mo); Arm 2:18 months (± 2 mo)), and Follow-up 3 (Arm 1:24 months (± 2 mo); Arm 2:30 months (± 2 mo))
Measure: Mean (Full Range); unit: scores on a scale
Groups:
- Arm 1: IMRT to Temporary Expander: Physical examination by MD, optional Breast MRI, Breast-Q© at baseline (after permanent implant exchange, physical exam and Breast-Q© may be done after the initiation of IMRT), 12 ± 2 months and 24 ± 2 months post- IMRT. Total length of the follow-up time will be 24 ± 2 months post-IMRT. A subset of 10 left-sided patients will receive 13N-NH3 PET scans within the radiation simulation session. A CT for coronary calcium scoring and a low-dose CT for attenuation correction will also be obtained at this time. Myocardial blood flow will be measured during rest and at peak stress with 13N-NH3 as a perfusion tracer. A follow-up 13N-NH3 PET study with low-dose CT for attenuation correction will be obtained 12-18 months (± 6 months) post-IMRT.
  Breast MRI
  Breast-Q© questionnaire
  Multi-Beam IMRT: The radiation dose (50-50.4 Gy/25-28 fractions in approximately 5-6 weeks), treatment-planning and delivery aspects are according to departmental guidelines for breast IMRT.
- Arm 2: IMRT to Permanent Implant: Physical examination by MD, optional Breast MRI, Breast-Q © at baseline (after permanent implant exchange and after IMRT), 18 ± 2 months and 30 ± 2 months post-IMRT, as these patients will undergo exchange of the temporary expander for the permanent implant approximately 4-8 months following the completion of radiation (at the discretion of the treating plastic surgeon). Total length of the follow-up time will be 30 ± 2 months post-IMRT
  Breast MRI
  Breast-Q© questionnaire
  Multi-Beam IMRT: The radiation dose (50-50.4 Gy/25-28 fractions in approximately 5-6 weeks), treatment-planning and delivery aspects are according to departmental guidelines for breast IMRT.
Arm/Group | Arm 1: IMRT to Temporary Expander | Arm 2: IMRT to Permanent Implant
Number analyzed (Participants) | 42 | 58
scores on a scale
  Baseline Physical Well Being Abdomen | 84 [76 to 92] | 64 [59 to 92]
  Follow-up 1 Physical Well Being Abdomen-Arm 1:12 months (± 2 mo); Arm 2:12-18 months (± 6 mo) | 70 [53 to 74] | 59 [47 to 70]
  Follow-up 2 Physical Well Being Abdomen-Arm 1:12-18 months (± 6 mo); Arm 2:18 months (± 2 mo) | 76 [62 to 79] | 69 [46 to 82]
  Follow-up 3 Physical Well Being Abdomen-Arm 1:24 months (± 2 mo); Arm 2:30 months (± 2 mo) | 69 [45 to 72] | 50 [0 to 75]
  Baseline Physical Well Being Chest | 68 [58 to 83] | 60 [55 to 67]
  Follow-up 1 Physical Well Being Chest-Arm 1:12 months (± 2 mo); Arm 2:12-18 months (± 6 mo) | 61 [50 to 74] | 63 [53 to 84]
  Follow-up 2 Physical Well Being Chest-Arm 1:12-18 months (± 6 mo); Arm 2:18 months (± 2 mo) | 66 [57 to 85] | 72 [58 to 81]
  Follow-up 3 Physical Well Being Chest-Arm 1:24 months (± 2 mo); Arm 2:30 months (± 2 mo) | 68 [50 to 88] | 68 [60 to 92]
  Baseline Psychosocial Well Being | 63 [50 to 67] | 67 [52 to 84]
  Follow-up 1 Psychosocial Well Being-Arm 1:12 months (± 2 mo); Arm 2:12-18 months (± 6 mo) | 63 [53 to 82] | 67 [50 to 86]
  Follow-up 2 Psychosocial Well Being-Arm 1:12-18 months (± 6 mo); Arm 2:18 months (± 2 mo) | 63 [52 to 70] | 63 [48 to 77]
  Follow-up 3 Psychosocial Well Being-Arm 1:24 months (± 2 mo); Arm 2:30 months (± 2 mo) | 62 [50 to 68] | 70 [52 to 100]
  Baseline Satisfaction with Breasts | 58 [52 to 66] | 52 [42 to 62]
  Follow-up 1 Satisfaction with Breasts-Arm 1:12 months (± 2 mo); Arm 2:12-18 months (± 6 mo) | 59 [48 to 79] | 59 [48 to 79]
  Follow-up 2 Satisfaction with Breasts-Arm 1:12-18 months (± 6 mo); Arm 2:18 months (± 2 mo) | 52 [44 to 73] | 48 [40 to 74]
  Follow-up 3 Satisfaction with Breasts-Arm 1:24 months (± 2 mo); Arm 2:30 months (± 2 mo) | 50 [43 to 60] | 58 [39 to 78]
  Baseline Satisfaction with Outcome | 67 [60 to 69] | 67 [47 to 75]
  Follow-up 1 Satisfaction with Outcome-Arm 1:12 months (± 2 mo); Arm 2:12-18 months (± 6 mo) | 67 [50 to 75] | 67 [57 to 75]
  Follow-up 2 Satisfaction with Outcome-Arm 1:12-18 months (± 6 mo); Arm 2:18 months (± 2 mo) | 61 [47 to 75] | 61 [47 to 75]
  Follow-up 3 Satisfaction with Outcome-Arm 1:24 months (± 2 mo); Arm 2:30 months (± 2 mo) | 0 [0 to 0] | 55 [40 to 70]
  Baseline Sexual Well Being | 51 [46 to 56] | 43 [34 to 55]
  Follow-up 1 Sexual Well Being-Arm 1:12 months (± 2 mo); Arm 2:12-18 months (± 6 mo) | 45 [36 to 52] | 47 [38 to 52]
  Follow-up 2 Sexual Well Being-Arm 1:12-18 months (± 6 mo); Arm 2:18 months (± 2 mo) | 45 [37 to 52] | 39 [32 to 60]
  Follow-up 3 Sexual Well Being-Arm 1:24 months (± 2 mo); Arm 2:30 months (± 2 mo) | 41 [27 to 50] | 48 [27 to 66]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | IMRT to Temporary Expander | IMRT to Permanent Implant
All-Cause Mortality (participants affected / at risk) | 0/42 | 8/58
Serious Adverse Events (participants affected / at risk) | 3/42 | 15/58
Other Adverse Events (participants affected / at risk) | 32/42 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT to Temporary Expander (N=42) | IMRT to Permanent Implant (N=58)
Breast infection (Infections and infestations) | 1 | 7
Breast pain (Reproductive system and breast disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wound infection (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT to Temporary Expander (N=42) | IMRT to Permanent Implant (N=58)
Alanine aminotransferase increased (Investigations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 6
Blood bilirubin increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 23 | 33
Neutrophil count decreased (Investigations) | 2 | 7
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 1
White blood cell decreased (Investigations) | 7 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT02086578/Prot_SAP_000.pdf